CLINICAL TRIAL: NCT03594773
Title: Dyadic Behavior Informatics for Psychotherapy Process and Outcome
Brief Title: Modeling Multi-level Dyadic Behavior to Transform the Science and Practice of Psychotherapy Process and Outcome.
Acronym: DAPPeR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Jeffrey Cohn, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO17110528; 171722822 (Other Grant/Funding Number: National Science Foundation)
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-06

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy; Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interpersonal Psychotherapy (Experimental): Participants randomized to this arm will be treated with 8 sessions over the course of 8 to 12 weeks by a therapist trained in IPT. Participants will complete brief questionnaires before and after treatment sessions. Before each session, they will report on their psychological distress. Following each session, participants and therapists will both complete assessments of the working alliance and rate their own and the other person's affective and interpersonal behavior.
  Interventions: Behavioral: Interpersonal Psychotherapy
- Cognitive Behavioral Therapy (Experimental): Participants randomized to this arm will be treated with 8 sessions over the course of 8 to 12 weeks by a therapist trained in CBT. Participants will complete brief questionnaires before and after treatment sessions. Before each session, they will report on their psychological distress. Following each session, participants and therapists will both complete assessments of the working alliance and rate their own and the other person's affective and interpersonal behavior.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will receive 8 one-on-one sessions over 8 to 12 weeks.
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Interpersonal Psychotherapy — Participants will receive 8 one-on-one sessions over 8 to 12 weeks.
  Other Names: IPT
  Arms: Interpersonal Psychotherapy

SUMMARY:
This is a short-term longitudinal study of psychotherapy process. Participants will be treated with 8 sessions of psychotherapy over the course of 8 to 12 weeks.

DETAILED DESCRIPTION:
Enrolled participants were randomized to one of two psychotherapy conditions: 8 sessions of Brief Cognitive Behavior Therapy or Brief Interpersonal Psychotherapy (IPT) over a 12 week protocol.

In response to the COVID-19 pandemic, we completed the study in two phases. Phase 1 procedures were conducted entirely in-person and Phase 2 procedures were conducted via telehealth. Phase 1 recruitment began July 2018 and concluded in February 2020. Recruitment for Phase 2 began July 2020 and concluded March 2021.

This project aims to model the dynamics of individual and dyadic behavior on a moment-by-moment basis within each therapy session and over the course of treatment. These models will be used to test hypotheses about multimodal behavior dynamics, psychotherapy process, type of treatment, and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65
2. Meet DSM-5 criteria for major depressive disorder (MDD), current episode, based on the Mini International Neuropsychiatric Interview (MINI)
3. Hamilton Rating Scale for Depression (HRSD-17) score ≥ 14 consistent with at least moderate depressive symptoms
4. If currently on antidepressant medication, must be on a stable dose for at least one month at the time of study entry and agree to remain on that dose for study duration
5. Fluent in English
6. Capacity to understand and give informed consent

Exclusion Criteria:

1. At high risk for suicide, that, in the clinical opinion of the investigator, would warrant a higher level of care such as hospitalization or intensive outpatient programs
2. Current depressive episode has psychotic features
3. Current depressive episode has been present for > 104 weeks
4. Meets criteria for substance use disorders, as defined by DSM-5, in the past 3 months, except for caffeine or nicotine. (Limited substance use, not meeting criteria for substance use disorders, is not exclusionary).
5. Meets DSM-5 criteria for prior manic or hypomanic episode (bipolar I or II disorder) or a psychotic disorder including schizoaffective disorder or schizophrenia
6. Meets DSM-5 criteria for antisocial personality disorder (MINI)
7. Significant, unstable, psychiatric co-morbidity that, in the opinion of the investigators, requires an alternative treatment approach (i.e., unstable eating disorder, unstable borderline personality disorder)
8. Significant unstable medical illness that may explain depressive symptoms such as epilepsy, autoimmune disorder, chronic pain, or unstable endocrine disorder
9. Cognitive deficits that would preclude completion of study questionnaires or participation in psychotherapy
10. Unable to unwilling to comply with study requirements (i.e., complete forms, attend sessions)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2018-07-08 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Cohn, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- WPIC/ Bellefield Towers/Depression and Manic Depression Prevention Program, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Swartz HA, Bylsma LM, Fournier JC, Girard JM, Spotts C, Cohn JF, Morency LP. Randomized trial of brief interpersonal psychotherapy and cognitive behavioral therapy for depression delivered both in-person and by telehealth. J Affect Disord. 2023 Jul 15;333:543-552. doi: 10.1016/j.jad.2023.04.092. Epub 2023 Apr 28. PMID 37121279
- [Derived] Girard JM, Yermol DA, Bylsma LM, Cohn JF, Fournier JC, Morency LP, Swartz HA. Dynamic and dyadic relationships between facial behavior, working alliance, and treatment outcomes during depression therapy. J Consult Clin Psychol. 2025 Nov;93(11):749-760. doi: 10.1037/ccp0000980. PMID 41182707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1 recruitment (in person delivery) began July 2018 and concluded in February 2020. Recruitment for Phase 2 (telehealth delivery) began July 2020 and concluded March 2021. Phase 2 recruitment: Phase 2 procedures was conducted virtually via Zoom to comply with COVID safety protocols. Recruitment took place at the University of Pittsburgh Medical Center using the Pitt+Me research registry.
Pre-assignment Details: No enrolled participants were excluded from the study prior to assignment to group as the assignment was done at the time of enrollment. Some participants were enrolled and assigned to a group but participated in no therapy sessions (lost to follow-up). Thus, the final numbers included in data analysis are slightly smaller than the total number initially enrolled.
Groups:
- Interpersonal Psychotherapy (IPT): Participants randomized to this arm will be treated with 8 sessions over the course of 8 to 12 weeks by a therapist trained in interpersonal psychotherapy (IPT). Participants will complete brief questionnaires before and after treatment sessions. Before each session, they will report on their psychological distress. Following each session, participants and therapists will both complete assessments of the working alliance and rate their own and the other person's affective and interpersonal behavior.
- Cognitive Behavioral Therapy (CBT): Participants randomized to this arm will be treated with 8 sessions over the course of 8 to 12 weeks by a therapist trained in cognitive-behavioral therapy (CBT). Participants will complete brief questionnaires before and after treatment sessions. Before each session, they will report on their psychological distress. Following each session, participants and therapists will both complete assessments of the working alliance and rate their own and the other person's affective and interpersonal behavior.
Period: Overall Study
Arm/Group | Interpersonal Psychotherapy (IPT) | Cognitive Behavioral Therapy (CBT)
Started (enrolled, randomized, and completed baseline assessment) | 42 | 35 (enrolled, randomized, and completed baseline assessment)
Completed (completed at least 1 session of intervention) | 36 | 29 (completed at least 1 session of intervention)
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Population: 77 participants completed the baseline assessment
Groups:
- Interpersonal Psychotherapy (IPT): Participants randomized to this arm will be treated with 8 sessions over the course of 8 to 12 weeks by a therapist trained in IPT. Participants will complete brief questionnaires before and after treatment sessions. Before each session, they will report on their psychological distress. Following each session, participants and therapists will both complete assessments of the working alliance and rate their own and the other person's affective and interpersonal behavior.
  Interpersonal Psychotherapy: Participants will receive 8 one-on-one sessions over 8 to 12 weeks.
- Cognitive Behavioral Therapy (CBT): Participants randomized to this arm will be treated with 8 sessions over the course of 8 to 12 weeks by a therapist trained in CBT. Participants will complete brief questionnaires before and after treatment sessions. Before each session, they will report on their psychological distress. Following each session, participants and therapists will both complete assessments of the working alliance and rate their own and the other person's affective and interpersonal behavior.
  Cognitive Behavioral Therapy: Participants will receive 8 one-on-one sessions over 8 to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Interpersonal Psychotherapy (IPT) | Cognitive Behavioral Therapy (CBT) | Total
Number analyzed (Participants) | 42 | 35 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] — age: continuous
  years | 32.10 (14.11) | 31.89 (13.23) | 32.0 (13.6)
Sex/Gender, Customized [Count of Participants; unit: Participants] — gender identity is categorical: male, female, other
  Participants
    Gender: Female | 25 | 26 | 51
    Gender: Male | 14 | 8 | 22
    Gender: Other | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 29 | 24 | 53
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 2 | 2
Hamilton Rating Scale for Depression - 17 [Mean (Standard Deviation); unit: units on a scale] — Our primary outcome measure of depression symptom severity was based on the Hamilton Rating Scale for Depression (HRSD-17) obtained at the final study visit (12 weeks). The HRSD-17 consists of 17 items with Likert scale of either 0 to 4 or 0 to 2. Total scores can range from 0(min) to 54(max), with higher scores indicating higher depression symptoms. Clinical interpretation of scale ranges of the HRSD-17 are as follows: 0-7= Normal 8-13= Mild Depression 14-18= Moderate Depression 19-22= Severe Depression >=23 = Very Severe Depression
  units on a scale | 19.51 (3.63) | 18.23 (3.17) | 18.92 (3.46)

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity
Description: Our primary outcome measure of depression symptom severity was based on the Hamilton Rating Scale for Depression (HRSD-17) obtained at the final study visit (12 weeks). The HRSD-17 consists of 17 items with Likert scale of either 0 to 4 or 0 to 2. Scores can range from 0(min) to 54(max), with higher scores indicating higher depression symptoms.
  Clinical interpretation of scale ranges of the HRSD-17 are as follows:
  0-7= Normal 8-13= Mild Depression 14-18= Moderate Depression 19-22= Severe Depression >=23 = Very Severe Depression
Time Frame: 12 weeks
Population: These analyses only include those who completed the final 12-week post-treatment assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interpersonal Psychotherapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 31 | 27
score on a scale | 11.9 (6.34) | 11.41 (5.41)
Statistical Analysis 1: Comparison: Interpersonal Psychotherapy vs Cognitive Behavioral Therapy; Test type: Superiority; p = .752, t-test, 2 sided; df=56, equal variances assumed; Mean Difference (Final Values) = -.496, 95% CI 2-sided [-3.62 to 2.63], Standard Error of Mean 1.56

2. Secondary Outcome: Working Alliance Inventory--Short Revised Client Version (WAI-SR-C)
Description: The Working Alliance Inventory-Short Revised (WAI-SR), client version, is a 12-item scale that measures three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Each subscale score for the WAI-SR ranges from 5(min) to 20(max), for a total score range of 15(min) to 60(max). Higher scores represent better alliance. The secondary outcome measure is based on the WAI-SR mean of the total scores measured at the final therapy visit (visit 8).
Time Frame: 12 weeks
Population: These analyses only include those who completed the WAI measure at all 8 treatment sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interpersonal Psychotherapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 27 | 24
score on a scale | 50.07 (8.08) | 51.33 (10.59)
Statistical Analysis 1: Comparison: Interpersonal Psychotherapy vs Cognitive Behavioral Therapy; Test type: Superiority; p = .633, t-test, 2 sided; df=49, equal variances assumed; Mean Difference (Final Values) = 1.26, 95% CI 2-sided [-4.01 to 6.52], Standard Error of Mean 2.62

3. Secondary Outcome: Working Alliance Inventory--Short Revised Therapist Version (WAI-SRT)
Description: The Working Alliance Inventory-Short Revised (WAI-SRT), therapist version, is a 12-item scale that measures three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of an affective bond. Each subscale score for the WAI-SR ranges from 5(min) to 20(max), for a total score range of 15(min) to 60(max). Higher scores represent better alliance. The secondary outcome measure is based on the WAI-SRT mean of the total scores measured at the final therapy visit (visit 8).
Time Frame: 12 weeks
Population: These analyses only include those who completed the WAI measure at all 8 treatment sessions.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Interpersonal Psychotherapy | Cognitive Behavioral Therapy
Number analyzed (Participants) | 28 | 23
score on a scale | 42.57 (5.83) | 43.52 (6.55)
Statistical Analysis 1: Comparison: Interpersonal Psychotherapy vs Cognitive Behavioral Therapy; Test type: Superiority; p = .586, t-test, 2 sided; df=49, equal variances assumed; Mean Difference (Final Values) = .950, 95% CI 2-sided [-2.53 to 4.44], Standard Error of Mean 1.73

ADVERSE EVENTS:
Time Frame: 12 weeks per participant
Arm/Group | Interpersonal Psychotherapy | Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/35
Other Adverse Events (participants affected / at risk) | 0/42 | 0/35

LIMITATIONS AND CAVEATS:
Limitations include the small sample size for each group and COVID-19 pandemic related restrictions necessitated that we conduct the 2nd half of the study virtually: delivery format for both intervention groups consisted of in person for the first phase of the trial (N=49) and virtual for the second phase of the trial (N=26). One participant for CBT and 3 for IPT were active in the study at the time of pandemic lockdown and had to be discontinued because of COVID-19 related safety requirements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT03594773/Prot_SAP_000.pdf